CLINICAL TRIAL: NCT03622606
Title: Development and Validation of a Language Screening Test in Acute Right Hemispheric Strokes
Acronym: R-LAST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Collaborators: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Principal Investigator, Dr Constance FLAMAND-ROZE, Neurosciences doctor, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P17/07_R-LAST
Record Dates: First submitted 2018-07-02; First posted 2018-08-09 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-03

CONDITIONS: Stroke
Keywords: Right hemispheric Stroke; Crossed aphasia; Acute phase
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute and subacute phase of right stroke (Experimental): The intervention will be the passation of Right Language Screening Test (R-LAST).
  Patients in acute phase of right hemispheric stroke will be used for the internal validation and the integrated reliability of the Right Language screening test.
  Patients in subacute phase of right hemispheric stroke will be used for the external validation of the Right Language screening test.
  Interventions: Diagnostic Test: Right Language screening test (R-LAST)

INTERVENTIONS:
Diagnostic Test: Right Language screening test (R-LAST) — Validation of the Right Language screening test in acute and subacute phase of right stroke

SUMMARY:
This is a bi-centric study whose main objective is the validation of a rapid screening test for language disorders in the acute phase of right hemisphere stroke.

Primary objective

The main objective is the validation of a rapid language disorder screening tool that will be used in the acute phase of right hemispheric stroke.

Secondary objectives

Secondary objectives are:

* Characterize the "atypical crossed aphasia" since the acute phase of stroke with a large cohort of patients , which, to our knowledge, has never been done.
* Re-evaluate the number of patients with acute language disorder in right hemisphere stroke.
* Validate the use of R-LAST by different categories of carers

DETAILED DESCRIPTION:
The R-LAST (Right Language screening test) comprises 8 subtests and a total of 15 items.

Validation will focus on the internal validity (no ceiling or floor effect, no redundancy, internal consistency), the external validity (against a "gold standard" in order to evaluate its specificity and its sensitivity) and the interclass agreement of R-LAST. The median time to administrate de scale will be calculated.

The investigators will validate the scale by administering it to 300 consecutive patients within 24 hours after admission to our 2 stroke units (Centre Hospitalier de Versailles and Centre hospitalier du sud francilien) and to 100 stabilized patients with and without atypical crossed aphasia using the MEC-P evaluation as a reference.

Patients must be 100% right-handed (Edinburgh test), be of French mother tongue, have no history of neurological disease, have no sensory disturbances (blindness, deafness) and no mirror crossed aphasia detected by the LAST (minimum score of 14/15 with a loss point granted for the "automatic speech" subtest, potentially stranded in right strokes)

ELIGIBILITY:
Inclusion Criteria:

* patients must be the age of majority
* Patients with right hemispheric stroke in the acute phase (internal validation + inter-examiner validation) or stabilization phase (external validation) confirmed by MRI or CT when MRI contraindicated
* Patient with no "mirror" crossed aphasia detected by the LAST procedure (A or B): LAST> 14
* Patients who read the newsletter
* Affiliation to a social security scheme

Criteria Exclusion:

* Minor patients
* No French speakers
* Patients with a history of stroke
* Patients with dementia
* Patients with sensory impairment: deafness, blindness
* Patient not 100% right handed in the Edinburgh questionnaire
* Inability to answer the Edinburgh Laterality Questionnaire and absence of any person to fill in the questionnaire.
* Patient with a left-handed person in its family
* Illiterate patients
* Patient presenting a "mirror" crossed aphasia detected by LAST A or B (score tolerated: 14/15 with error accepted to the automatic speech)
* Inability to receive the information letter about the protocol and to read the newsletter
* Refusal of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-09-25 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Score at R-LAST | Day 1
  Internal validation: no item will present effect floor, ceiling or of redundancy.
  Validation inter examiner: the score obtained to R-LAST is independent from the examiner.
  External validation: the patients detected by gold standard as presenting a speech difficulty bound to a right hemispherical lesion will also be him by R-LAST (no forgery negatives), and that the patients not presenting speech difficulty during the signing of these standard gold will obtain the maximum score to R-LAST (no forgery positive).

SECONDARY OUTCOMES:
Score at LAST A and B | Day 1
  Detect the patients presenting a right hemispherical AVC with crossed aphasia "mirror"
Time of signing R-LAST | Day 1
  To obtain an average time of signing which will have to be shorter than that of the standard gold used during the external validation.
Simplicity and convenience of R-LAST | Day 1
  Contains only a sheet printed in black and white and both sides (to avoid the semantic indications bound to the color of an item, and to simplify the reproduction).
Visual aspect of R-LAST | Day 1
  Presentation in "portrait" mode, so that patients presenting a neurovisual disorder of type héminégligence or héminanopsie controlatérale are not penalized

CONTACTS AND LOCATIONS:
Overall Officials: Didier SMADJA, Neurologist, Principal Investigator — Sud Francilien Hospital
Locations (2):
- France (2):
  - CH Sud Francilien, Corbeil-Essonnes
  - CH de Versailles, Le Chesnay

IPD SHARING:
Plan to Share IPD: Undecided